CLINICAL TRIAL: NCT06433947
Title: A Phase 1b, Dose Escalation/Dose Expansion, Multicenter, Open-Label Study to Assess the Safety and Tolerability of OPN-6602 Monotherapy and in Combination With Dexamethasone in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Study to Assess Safety and Tolerability of OPN-6602 in Subjects With Relapsed and/or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Opna Bio LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPN6602-C01
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation monotherapy (Experimental)
  Interventions: Drug: OPN-6602
- Dose escalation in combo with dexamethasone (Experimental)
  Interventions: Drug: OPN-6602; Drug: Dexamethasone
- Dose expansion (Experimental)
  Interventions: Drug: OPN-6602

INTERVENTIONS:
Drug: OPN-6602 — orally active, small molecule inhibitor of EP300 and CBP bromodomain; dosed daily
Drug: Dexamethasone — Synthetic glucocorticoid; 40 mg Days 1, 8, 15 of each cycle
  Arms: Dose escalation in combo with dexamethasone

SUMMARY:
Phase 1b, open-label study evaluating the safety, tolerability, pharmacokinetics, preliminary antitumor activity, and pharmacodynamics of OPN-6602 monotherapy and in combination with dexamethasone in subjects with relapsed and/or refractory MM.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma (MM)
* Relapsed or refractory to 3 or more different prior lines of therapy for MM that included immunomodulatory agents, proteosome inhibitors, and anti-CD38 antibody and not a candidate for or intolerant to established therapy known to provide clinical benefit
* Adequate hematologic, renal, liver, cardiac function

Exclusion Criteria:

* Monoclonal gammopathy of undetermined significance (MGUS), smoldering myeloma, Waldenström's macroglobulinemia, or IgM myeloma
* Active plasma cell leukemia
* Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes (POEMS syndrome)
* Prior Stevens Johnson syndrome
* Localized radiation therapy to disease site(s) within 2 weeks of the first dose
* Prior autologous peripheral stem cell transplant or prior autologous bone marrow transplantation within <90 days of the first dose of study drug
* Prior allogeneic stem cell transplantation or solid organ transplantation within 12 months of screening; subjects receiving immunosuppressive medication for active graft vs host disease will be excluded.
* Prior chemotherapy, targeted anticancer or radiation therapy within 2 weeks prior to first dose of study drug
* Concomitant high-dose corticosteroids (except subjects on chronic steroids given for disorders other than myeloma)
* Known central nervous system involvement by multiple myeloma
* Active known second malignancy with exception of adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer; adequately treated Stage 1 cancer from which the subject is currently in remission and has been in remission for ≥2 years; low-risk prostate cancer with a Gleason score <7 and a PSA level <10 ng/mL; any other cancer from which the subject has been disease-free for ≥3 years
* Ongoing systemic infection requiring parenteral treatment
* Poorly controlled Type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number and type of dose-limiting toxicities (DLTs) | Through up to approximately 30 days following last dose of OPN-6602
Number and type of treatment-emergent adverse events (TEAEs) | Through up to approximately 30 days following last dose of OPN-6602
Number of Participants With Clinical Laboratory Test Abnormalities | Through up to approximately 30 days following last dose of OPN-6602
  Number of participants who experienced a clinical laboratory test abnormality, including hematology and serum chemistry, and coagulation. Abnormalities considered are those Grade 3-4 events with a >= 1 grade increase from baseline using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Banner MD Anderson, Gilbert, Arizona
  - Stanford Cancer Institute, Stanford, California
  - Emory Winchip Cancer Center, Atlanta, Georgia
  - University of Kansas Clinical Research Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - Huntsman Cancer Center Institute University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No